CLINICAL TRIAL: NCT07246746
Title: Use of an Infotainment System in MRI in Patients Suffering From Unexpected Anxiety.
Acronym: USIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MIGNOT AOIparaM 2023
Record Dates: First submitted 2025-09-26; First posted 2025-11-24 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Unexpected Anxiety
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Innovision© (Experimental)
  Interventions: Other: Assessment of patient anxiety through self-administration of the State Anxiety Inventory Form Y-A questionnaire; Other: Anxiety support procedure according to randomization: Innovision© or Hypnosis
- Hypnosis control (Active Comparator)
  Interventions: Other: Assessment of patient anxiety through self-administration of the State Anxiety Inventory Form Y-A questionnaire; Other: Anxiety support procedure according to randomization: Innovision© or Hypnosis

INTERVENTIONS:
Other: Assessment of patient anxiety through self-administration of the State Anxiety Inventory Form Y-A questionnaire — Assessment of patient anxiety
Other: Anxiety support procedure according to randomization: Innovision© or Hypnosis — Hypnosis or Innovision device

SUMMARY:
MRI scans are now considered essential for diagnosing or monitoring disease, and as a result, the number of MRI scans has increased significantly in recent years.

Nevertheless, these routine examinations remain a source of apprehension and anxiety for some people.

The objective of this study is to compare two methods of care, enabling anxious individuals to complete their MRI examination and obtain images of sufficient quality for the radiologist to read and interpret.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have given their verbal consent
* Individuals over the age of 18
* Hospitalized or ambulatory individuals who are able-bodied and scheduled to undergo a brain MRI scan on the 1.5T A MRI machine at the Dijon University Hospital.
* Individuals reporting anxiety about brain MRI for the first time upon admission by the radiology technician.

Exclusion Criteria:

* Persons not affiliated with or not covered by a social security system
* Persons subject to legal protection measures (guardianship, trusteeship)
* Persons subject to judicial protection measures
* Women who know they are pregnant
* Adults who are incapable or unable to give their consent
* Persons with contraindications to MRI
* Persons who have already undergone an MRI accompanied by hypnosis
* Persons who do not speak French
* Persons who cannot read French
* Persons with cognitive disorders
* Persons who have taken sedatives before the examination
* Persons who regularly take anxiolytic medication and have increased their usual dose before the examination
* Persons who have already participated in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of brain MRI sequences reported as interpretable | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France